CLINICAL TRIAL: NCT04102826
Title: Personalised Approach to Restoration of Arm Function in People With High-level Tetraplegia
Brief Title: Restoration of Arm Function in People With High-level Tetraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Collaborators: Engineering and Physical Sciences Research Council, UK (Other); Keele University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: RobertJAH
Record Dates: First submitted 2019-09-09; First posted 2019-09-25 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Incomplete Spinal Cord Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Functional electrical stimulation (FES) — Functional electrical stimulation combined with mobile arm support to restore upper limb function.

SUMMARY:
Functional electrical stimulation (FES) has been used to activate paralysed muscles and restore movement after spinal cord injury and stroke. This technology involves the application of low-level electrical currents to the nerves and muscles to cause muscle contraction where the user's ability to achieve that through voluntary means has been lost.

Providing control of muscle contraction in a coordinated way can mean that users are able once again to produce functional movements in otherwise paralysed limbs.

Routine clinical use is limited to the prevention of drop foot in the lower limb following stroke and occasional therapeutic use in the hand and shoulder. Systems providing functional reach and grasp, however, have not achieved clinical or commercial success. This project aims to develop methods for personalising assistive technology to restore arm function in people with high-level spinal cord injury. The investigators will use a combination of electrical stimulation to elicit forces in muscles no longer under voluntary control, and mobile arm supports to compensate for insufficient muscle force where necessary. The investigators will use computational models specific to an individual's functional limitations to produce patient-specific interventions. The project will be in three phases: building a model to predict the effects of electrical stimulation on a paralysed arm with arm support, development of methodologies using this model to optimise the arm support and stimulation system, and testing of stimulation controllers designed using this approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mid- to high-level spinal cord injury resulting in partial or full paralysis of the upper limb will be eligible for inclusion in the study. In addition, they must be:
* Able to give informed consent;
* Able to remain comfortably seated with provision of trunk stability;
* Medically stable and at least six weeks from injury; and
* Have sufficient passive range of motion without discomfort.

Exclusion Criteria:

* Have orthopaedic implants across or between electrode sites;
* Have active cardiac implant;
* Have poor skin conditions, scar or carcinogenic tissue at site of stimulation;
* Have uncontrolled pain;
* Have uncontrolled epilepsy;
* Have skin reactions to electrodes;
* Have open wounds or injuries; and
* Are pregnant or planning for a pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Change in Canadian Occupational Performance Measure (COPM) | At baseline and at study completion for each participant. Study completion will be up to 6 months after the baseline measurement.
  The COPM is a questionnaire based assessment of performance and satisfaction of functional tasks. The COPM measures an individuals self-perception of occupational performance over time. This is a 10 point scale, with 1 indicating poor performance and low satisfaction, and 10 indicating very good performance and high satisfaction. The scale is applied to up to 5 problems identified by an individual that affect their everyday life. An average score is then calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Postans, PhD, Principal Investigator — RJAH Orthopaedic Hospital NHS Foundation Trust
Locations (1):
- Neil Postans, Oswestry, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No